CLINICAL TRIAL: NCT05839028
Title: Mechanisms of Left Ventricular Remodeling in Hypertensive Patients Working on a Rotational Expeditionary Basis in the Conditions of the Arctic Region
Brief Title: Mechanisms of LV Remodeling in Hypertensive Patients Working on a Rotational Expeditionary Basis in the Arctic
Status: Active, not recruiting | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: TomskNRMC HD
Record Dates: First submitted 2023-04-05; First posted 2023-05-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: hypertension; Arctic; rotational shift work; echocardiography
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Biomarkers of inflammation and biomarkers that allow to detect heart failure with preserved ejection fraction at an early stage
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with hypertension of stages 1 and 2: Individuals with stage 1 and 2 hypertension living in a temperate climate zone and doing rotational shiftwork in the Arctic.
- Healthy volunteers: Virtually healthy individuals living in a temperate climate zone and and doing rotational shiftwork in the Arctic.

SUMMARY:
The main goal of our investigation is to study the mechanisms of formation of left ventricular remodeling in patients with hypertension, working on a rotational expedition basis in the Arctic.

DETAILED DESCRIPTION:
Hypothesis: In patients with hypertension working in the conditions of the Arctic shift, the combination of climatic and geographical factors and rotational expeditionary method of labor contributes to the increase in the left ventricular remodeling processes and leads to the formation of heart failure with preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* The patient signed the informed consent

Exclusion Criteria:

* Valvular pathology of the heart
* Past cardiac or cerebral complications
* Identified heart rhythm disturbances
* Coronary heart disease
* Patients with severe somatic pathology, whose prognostic survival rate does not exceed 1 year
* The presence of a mental disorder of organic origin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Зatients with hypertension of stages 1 and 2 and practically healthy individuals living in a temperate climate zone and carrying out an Arctic watch. Hypertension in the Arctic is characterized by faster target organ damage and worse prognosis.
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic assessment of GLS (Global longitudinal strain), % | One year
  Echocardiographic assessment of global strain (%) at baseline and after one year of follow-up.

SECONDARY OUTCOMES:
Concentration of Myeloperoxidase, ug/mL | One year
  Concentration of oxidative stress biomarker, myeloperoxidase, is assessed using Lab analyzer Stat Fax 4200 (USA).
Concentration of oxidized low density lipoproteins, CU | One year
  Concentration of oxidative stress biomarker, oxidized low density lipoproteins, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of homocysteine, umol/L | One year
  Concentration of oxidative stress biomarker, homocysteine, is assessed using Lab analyzer - IMMULITE 2000 (Siemens Diagnostics, USA).
Concentration of C-reactive protein, IU/L | One year
  Concentration of immune inflammation biomarker, C-reactive protein, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of tumor necrosis factor alpha, pg/ml | One year
  Concentration of immune inflammation biomarker, tumor necrosis factor alpha is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of 1,6,8 interleukins, pg/mL | One year
  Concentration of immune inflammation biomarker, (1,6,8) interleukin, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of GDF-15/MIC-1 (Growth Differentiation Factor 15/Macrophage-inhibitory 1), pg/mL | One year
  Concentration fibrosis biomarker, GDF-15/MIC-1, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of PIIINP (N-terminal propeptide to procollagen III), ng/mL | One year
  Concentration of fibrosis biomarker, PIIINP, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of FGF-23 (Fibroblast growth factor 23), pmol/L | One year
  Concentration of fibrosis biomarker, FGF-23, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of plasma procollagen type 3, CU | One year
  Concentration of remodeling factor biomarker, plasma procollagen type 3, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of adrenaline, pg/mL | One year
  Concentration of catecholamine, adrenaline, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of noradrenaline, pg/mL | One year
  Concentration of catecholamine, noradrenaline, is assessed using Lab analyzer - Stat Fax 4200 (USA);
Concentration of testosterone, nmol/L | One year
  Concentration of hormone, testosterone, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of progesterone, nmol/L | One year
  Concentration of hormone biomarker, progesterone, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of estradiol, pg/mL | One year
  Concentration of hormone, estradiol, is assessed using Lab analyzer - Stat Fax 4200 (USA).
Concentration of cystatin-C, ng/mL | One year
  Concentration of chronic kidney disease biomarker, cystatin-C, is assessed by Lab analyzer - Stat Fax 4200 (USA).
Concentration of NGAL (Neutrophilic gelatinase-associated lipocalin or neutrophilic lipocalin), ng/mL | One year
  Concentration of chronic kidney disease biomarker, NGAL, is assessed by Lab analyzer - Stat Fax 4200 (USA).

CONTACTS AND LOCATIONS:
Overall Officials: Liudmila Gapon, MD, PhD, Principal Investigator — Tyumen Cardiology Research Center
Locations (1):
- Tyumen Cardiology Research Center, Tyumen, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data warehouse but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.